CLINICAL TRIAL: NCT05025124
Title: Entia Liberty: Analytical Performance Validation - Accuracy and Precision
Brief Title: Entia Liberty: Accuracy and Precision
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 304727
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Method comparison: 400 samples to be compared directly against the reference method. This is to get the bias estimate.
  Interventions: Device: Entia Liberty
- Precision: 30 samples will be each split into 10 individual samples to evaluate the precision of the Entia Liberty devices.
  Interventions: Device: Entia Liberty

INTERVENTIONS:
Device: Entia Liberty — Home monitoring system

SUMMARY:
This study forms part of Entia's clinical evidence for regulatory submission. This study evaluates Entia Liberty's performance claims with venous blood compared to the gold standard clinical laboratory haematology analysers. Excess blood flagged by the laboratory meeting our requirements will be tested on the Entia Liberty device and have its results compared against the laboratory results. Samples will also be flagged for precision testing (same blood sample, split into 10 Entia Liberty samples).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Currently receiving standard of care systemic anti-cancer therapy (chemotherapy, immunotherapy, endocrine and targeted therapy) for solid organ malignancy and has received at least one cycle
* Blood samples that have been stored in K2-EDTA vacutainers only
* For Accuracy testing: Samples covering 75% of parameter ranges (Neutrophils: 0.5-7.5 x 109/L, Platelets: 20-450 x 109/L, Haemoglobin: 70-180 g/L), These will be determined by a gold standard analyser which has been recently calibrated.
* Reliability study: Level range per parameter. These will be determined by a gold standard analyser which has been recently calibrated.
* Neutrophils (We assume WBC to behave similarly in the same ranges) Low: 0.5-1.2 x 109/L (3 samples), 1.2-2 x 109/L (2 samples) Normal: 2-7 x 109/L (3-4 samples) High: 7-12 x 109/L (1-2 samples)
* Platelets Low: 50-150 x 109/L (5 samples) Normal: 150-400 x 109/L (3 - 4 samples) High: >400 x 109/L (1-2 samples)
* Haemoglobin Low: <120 g/L (5 samples) Normal: 120-170 g/L (3 - 4 samples) High: >170 g/L (1-2 samples)

Exclusion Criteria:

* History of haematological malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No participants will be recruited. Samples used are from excess venous bloods from the Christie haematology laboratory
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
To obtain the Total Error per parameter from the results of the Entia Liberty device | 3 months
  The dataset from this study will provide evidence to support the device's performance claims.
To obtain the linearity per parameter from the results of the Entia Liberty device | 3 months
  The dataset from this study will provide evidence to support the device's performance claims.
To obtain the bias per parameter from the results of the Entia Liberty device | 3 months
  The dataset from this study will provide evidence to support the device's performance claims.
To obtain the precision per parameter from the results of the Entia Liberty device | 3 months
  The dataset from this study will provide evidence to support the device's performance claims.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom